CLINICAL TRIAL: NCT03004872
Title: Relationship Between Postpartum Mood Disorders and Delivery Experience
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Joanna Kountanis, Assistant Professor, University of Michigan
Other Study IDs: HUM00119428
Record Dates: First submitted 2016-11-15; First posted 2016-12-29 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Postpartum Period; Depression; Stress Disorders, Post-Traumatic
Keywords: birth experience; postpartum depression; PTSD; pain during labor; pain during cesarean delivery; non-elective induction of labor; unplanned surgery for urgent/emergent cesarean delivery; postpartum hemorrhage
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic; Depression, Postpartum; Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate potential risk factors for developing postpartum depression or posttraumatic stress disorder during the first year postpartum in patients who have no preexisting history of PTSD or PPD.

DETAILED DESCRIPTION:
It is theorized that poor pain control during labor and cesarean delivery, non-elective inductions, unplanned surgeries such as urgent/emergent cesarean delivery or operating room management of postpartum hemorrhage, and opioid abuse/addiction are risk factors for developing postpartum depression (PPD) or post-traumatic stress disorder (PTSD) after delivery. This study will, through questionnaires, interviews, and examination of the medical record, seek to identify whether and how strongly such correlations exist during the first year postpartum in patients who have no preexisting history of these conditions.

ELIGIBILITY:
Inclusion Criteria:

* Woman planning on giving birth at the University of Michigan
* Speaks English without translator
* Live pregnancy not desiring termination
* Smartphone owner
* Woman whose delivery date is >28 weeks gestational age

Exclusion Criteria:

* History of previous postpartum depression (PPD) or posttraumatic stress disorder (PTSD) from a birth experience
* Non-English speaker requiring a translator
* Patients who have a fetus with major fetal anomalies
* Positive screening at 28 weeks antepartum for Edinburgh Postnatal Depression Scale (EPDS) or Primary Care PTSD (PC-PTSD) screen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women who are planning to give birth at the University of Michigan.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Association of poor birth experiences with development of postpartum posttraumatic stress disorder (PTSD). | 1 year postpartum
  Enrollees will receive questionnaires for Perinatal Posttraumatic Stress Disorder (PPQ) screenings 6 weeks, 3 months, 6 months, and 1 year postpartum. Positive screens are defined as PPQ>19. PPQ>13 will be considered as subsyndromal. At each screening, patients with positive scores will be interviewed to diagnose PTSD and to look for thematic similarities in birth experiences. Patients' medical charts will be reviewed for 4 clinical events: Pain scores >5 with a labor epidural in place; Pain during cesarean delivery requiring general anesthesia, IV narcotics, ketamine, midazolam, nitrous oxide, or reassurance; Non-elective inductions of labor; and Unplanned surgery including urgent/emergent cesarean delivery and postpartum hemorrhage requiring operating room management. Statistical analysis of all 4 PPQ scores and evaluation of clinical birth events will be performed to determine the association of poor birth experiences with postpartum depression.
Association of poor birth experience with development of postpartum depression. | 1 year postpartum
  Enrollees will receive questionnaires for Edinburgh Postnatal Depression Scale (EPDS) screenings at 6 weeks, 3 months, 6 months, and 1 year postpartum. Positive screens are defined as EPDS score >10 or a positive response for question 10 asking about suicidality. At each screening, patients with positive scores will be interviewed to diagnose depression and to look for thematic similarities in birth experiences. Patients' medical charts will be reviewed for 4 clinical events: Pain scores >5 with a labor epidural in place; Pain during cesarean delivery requiring general anesthesia, IV narcotics, ketamine, midazolam, nitrous oxide, or reassurance; Non-elective inductions of labor; and Unplanned surgery including urgent/emergent cesarean delivery and postpartum hemorrhage requiring operating room management. Statistical analysis of all 4 EPDS scores and evaluation of clinical birth events will be performed to determine the association of poor birth experiences with postpartum depression.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Kountanis, MD, Principal Investigator — University of Michigan; Elizabeth Langen, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kountanis JA, Kirk R, Handelzalts JE, Jester JM, Kirk R, Muzik M. The associations of subjective appraisal of birth pain and provider-patient communication with postpartum-onset PTSD. Arch Womens Ment Health. 2022 Feb;25(1):171-180. doi: 10.1007/s00737-021-01154-z. Epub 2021 Jul 12. PMID 34250546